CLINICAL TRIAL: NCT05333289
Title: Phase 1/2, Randomized, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1020 and mRNA-1030 Candidate Seasonal Influenza Vaccines in Healthy Adults
Brief Title: A Study of mRNA-1020 and mRNA-1030 Seasonal Influenza Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1020-P101
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Seasonal Influenza
Keywords: Influenza vaccine; mRNA-1020; mRNA-1030; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- mRNA-1030 Dose Level A (Experimental): Participants will receive mRNA-1030 at Dose Level A by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1030
- mRNA-1020 Dose Level A (Experimental): Participants will receive mRNA-1020 at Dose Level A by IM injection on Day 1.
  Interventions: Biological: mRNA-1020
- mRNA-1030 Dose Level B (Experimental): Participants will receive mRNA-1030 at Dose Level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1030
- mRNA-1020 Dose Level B (Experimental): Participants will receive mRNA-1020 at Dose Level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1020
- mRNA-1030 Dose Level C (Experimental): Participants will receive mRNA-1030 at Dose Level C by IM injection on Day 1.
  Interventions: Biological: mRNA-1030
- mRNA-1020 Dose Level C (Experimental): Participants will receive mRNA-1020 at Dose Level C by IM injection on Day 1.
  Interventions: Biological: mRNA-1020
- mRNA-1010 (Active Comparator): Participants will receive mRNA-1010 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Active Comparator (Active Comparator): Participants will receive an active comparator by IM injection on Day 1.
  Interventions: Biological: Active Comparator

INTERVENTIONS:
Biological: mRNA-1030 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1030 Dose Level A; mRNA-1030 Dose Level B; mRNA-1030 Dose Level C
Biological: mRNA-1020 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1020 Dose Level A; mRNA-1020 Dose Level B; mRNA-1020 Dose Level C
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010
Biological: Active Comparator — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: Active Comparator

SUMMARY:
The primary objective of this study is to evaluate the safety, reactogenicity, and humoral immunogenicity of mRNA-1020, mRNA-1030, and mRNA-1010 vaccines against vaccine-matched influenza A and B strains.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 kilograms (kg)/square meter (m^2) to 35 kg/m^2 (inclusive) at the Screening Visit.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 90 days following vaccine administration, and not currently breastfeeding.

Exclusion Criteria:

* Participant has had close contact to someone with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or COVID-19 as defined by the Centers for Disease Control and Prevention (CDC) or has had a positive SARS-CoV-2 test in the past 10 days prior to the Screening Visit.
* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 180 days prior to screening (for corticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Participant has received or plans to receive any licensed or authorized vaccine, including COVID-19 vaccines, ≤28 days prior to the study injection (Day 1) or plans to receive a licensed or authorized vaccine within 28 days after the study injection.
* Participant has received a Northern Hemisphere (NH) 2021-2022 seasonal influenza vaccine or any other influenza vaccine within 180 days prior to Day 1.
* Participant tested positive for influenza by CDC-recommended testing methods within 180 days prior to Day 1.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Foothills Research Center, Phoenix, Arizona
  - Alliance for MultiSpecialty Research, Coral Gables, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - IACT Health, Columbus, Georgia
  - Meridian Clinical Research, Sioux City, Iowa
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, Endwell, New York
  - Lucas Research, Morehead City, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Meridian Clinical Research, Cincinnati, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - LinQ Research, LLC, Pearland, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - South Ogden Family Medicine, South Ogden, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Flublok: Participants received Flublock by intramuscular (IM) injection on Day 1.
- mRNA-1010: Participants received mRNA-1010 by IM injection on Day 1.
- mRNA-1030 Dose Level A: Participants received mRNA-1030 Dose Level A by IM injection on Day 1.
- mRNA-1020 Dose Level A: Participants received mRNA-1020 Dose Level A by IM injection on Day 1.
- mRNA-1030 Dose Level B: Participants received mRNA-1030 Dose Level B by IM injection on Day 1.
- mRNA-1020 Dose Level B: Participants received mRNA-1020 Dose Level B by IM injection on Day 1.
- mRNA-1030 Dose Level C: Participants received mRNA-1030 Dose Level C by IM injection on Day 1.
- mRNA-1020 Dose Level C: Participants received mRNA-1020 Dose Level C by IM injection on Day 1.
Period: Overall Study
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Started | 72 | 71 | 71 | 72 | 72 | 71 | 72 | 71
Received at Least 1 Dose of Investigational Product | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Safety Set (The Safety Set consisted of all randomly assigned participants who received the investigational product.) | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Solicited Safety Set (The Solicited Safety Set consisted of all participants in the Safety Set who contributed any solicited adverse reaction data.) | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Completed | 62 | 69 | 67 | 64 | 67 | 62 | 67 | 67
Not Completed | 10 | 2 | 4 | 8 | 5 | 9 | 5 | 4
Not completed — Other | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 1 | 6 | 3 | 3 | 2 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomization Set consisted of all participants who were randomly assigned.
Groups:
- Flublok: Participants received Flublock by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C | Total
Number analyzed (Participants) | 72 | 71 | 71 | 72 | 72 | 71 | 72 | 71 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (14.51) | 46.0 (15.03) | 47.1 (14.40) | 48.0 (16.50) | 46.9 (14.11) | 48.0 (14.84) | 47.3 (17.13) | 49.2 (15.88) | 47.4 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 44 | 42 | 38 | 41 | 39 | 40 | 314
  Male | 35 | 38 | 27 | 30 | 34 | 30 | 33 | 31 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 6 | 7 | 6 | 8 | 4 | 6 | 50
  Not Hispanic or Latino | 63 | 66 | 65 | 65 | 65 | 63 | 67 | 65 | 519
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 8
  Asian | 3 | 3 | 3 | 0 | 4 | 2 | 4 | 3 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 6 | 11 | 15 | 6 | 13 | 10 | 7 | 6 | 74
  White | 60 | 52 | 51 | 65 | 54 | 58 | 61 | 59 | 460
  More than one race | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in the electronic diary (eDiary). Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section and presented by each dose group separately.
Time Frame: Up to Day 7 (7 days after vaccination)
Population: The Solicited Safety Set consisted of all participants in the Safety Set who contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Participants
  Solicited Local ARs | 37 | 63 | 59 | 60 | 57 | 58 | 67 | 67
  Solicited Systemic ARs | 32 | 61 | 44 | 57 | 55 | 58 | 64 | 64

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent AE (TEAE) was defined as any event not present before exposure to vaccine or any event already present that worsens in intensity or frequency after exposure. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsens from baseline and is considered clinically significant in the medical and scientific judgment of the Investigator. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study, regardless of causality, is located in the "Reported Adverse Events" section and presented by each dose group separately.
Time Frame: Up to Day 28 (28 days after vaccination)
Population: The Safety Set consisted of all randomly assigned participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Participants | 10 | 17 | 6 | 15 | 11 | 15 | 12 | 21

3. Primary Outcome: Number of Participants With Medically-Attended AEs (MAAEs), Adverse Event of Special Interest (AESI), AEs Leading to Withdrawal and Serious Adverse Events (SAEs)
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that leads to an unscheduled visit to an healthcare practitioner. This would include visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or COVID-19 and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section and presented by each dose group separately.
Time Frame: Day 1 through Day 181
Population: The Safety Set consisted of all randomly assigned participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 72 | 67 | 72 | 70
Participants
  Medically-Attended AEs | 23 | 20 | 16 | 24 | 18 | 19 | 17 | 23
  Adverse Event of Special Interest | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
  AEs Leading to Withdrawal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 4

4. Primary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29 as Measured by Hemagglutination Inhibition (HAI) Assay Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
Time Frame: Day 29
Population: PP Set consisted of all participants in the FAS who complied with injection schedule, complied with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, did not had influenza infection at baseline through Day 29, and had no major protocol deviations that impacted immune response. Number of participants analyzed signifies those who were evaluable for this outcome measure and number analyzed signifies those who were evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 65 | 61 | 67 | 63 | 63 | 60 | 66 | 61
titer
  Influenza A H1N1 Antibody | 724.69 [527.41 to 995.78] | 498.43 [392.33 to 633.22] | 328.44 [243.71 to 442.62] | 472.81 [345.73 to 646.61] | 387.92 [291.94 to 515.47] | 378.34 [267.06 to 535.99] | 431.61 [325.80 to 571.78] | 527.55 [404.11 to 688.70]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody | 354.11 [269.13 to 465.92] | 316.36 [243.84 to 410.45] | 239.78 [180.19 to 319.07] | 263.95 [206.13 to 338.00] | 211.86 [152.96 to 293.44] | 255.44 [181.20 to 360.09] | 283.59 [222.40 to 361.62] | 300.62 [228.60 to 395.34]
  Influenza B/Victoria Lineage | 151.68 [116.74 to 197.06] | 88.57 [69.14 to 113.47] | 86.86 [70.52 to 106.99] | 86.88 [68.90 to 109.55] | 105.92 [85.24 to 131.60] | 82.86 [64.68 to 106.13] | 91.71 [73.63 to 114.23] | 75.56 [58.47 to 97.65]
  Influenza B/Yamagata Lineage | 277.06 [225.13 to 340.96] | 245.01 [196.73 to 305.41] | 191.74 [157.35 to 233.65] | 249.81 [199.09 to 313.45] | 237.78 [194.08 to 291.31] | 246.78 [196.09 to 310.57] | 255.31 [216.23 to 301.44] | 243.62 [196.35 to 302.26]

5. Primary Outcome: GMT of Anti-Neuraminidase (NA) Antibodies at Day 29 as Measured by Neuraminidase Inhibition (NAI) Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
Time Frame: Day 29
Population: The Per Protocol (PP) Set consisted of all participants in the Full analysis set (FAS) who complied with injection schedule, complied with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, did not had influenza infection at baseline through Day 29, and had no major protocol deviations that impacted immune response. Here, Number analyzed signifies those who were evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 67 | 63 | 67 | 66 | 66 | 64 | 67 | 63
titer
  Influenza A H1N1 Antibody | 103.61 [91.50 to 117.33] | 97.52 [88.13 to 107.91] | 163.35 [134.09 to 198.99] | 219.26 [174.90 to 274.86] | 195.34 [159.57 to 239.11] | 198.70 [160.51 to 245.98] | 170.25 [141.09 to 205.43] | 268.35 [210.93 to 341.40]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 67 | 63 | 67 | 66 | 66 | 64 | 66 | 63
  Influenza A H3N2 Antibody | 20.49 [16.47 to 25.51] | 21.09 [16.44 to 27.05] | 69.21 [50.36 to 95.12] | 105.23 [78.54 to 141.00] | 79.56 [57.45 to 110.18] | 127.60 [92.74 to 175.55] | 92.57 [70.53 to 121.49] | 139.16 [104.11 to 186.00]
  Influenza B/Victoria Lineage | 69.93 [60.15 to 81.31] | 78.26 [66.50 to 92.10] | 268.39 [232.82 to 309.40] | 416.08 [354.45 to 488.42] | 316.66 [269.21 to 372.46] | 477.73 [402.55 to 566.95] | 316.71 [270.66 to 370.58] | 470.32 [390.92 to 565.83]
  Influenza B/Yamagata Lineage | 183.03 [146.21 to 229.13] | 215.34 [174.21 to 266.19] | 837.52 [718.85 to 975.80] | 1293.51 [1099.70 to 1521.48] | 953.89 [823.81 to 1104.52] | 1441.95 [1215.88 to 1710.05] | 998.57 [857.69 to 1162.59] | 1428.87 [1186.31 to 1721.02]

6. Primary Outcome: Geometric Mean Fold-Rise (GMFR) of Anti-HA Antibodies at Day 29 as Measured by HAI Assay Vaccine-Matched Seasonal Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI for GMFR was calculated based on the t distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 65 | 61 | 67 | 63 | 63 | 60 | 66 | 61
ratio
  Influenza A H1N1 Antibody | 9.93 [6.60 to 14.94] | 9.12 [6.63 to 12.55] | 5.29 [3.77 to 7.42] | 8.56 [6.03 to 12.15] | 6.83 [4.96 to 9.39] | 8.39 [5.93 to 11.88] | 6.73 [5.01 to 9.04] | 6.79 [4.86 to 9.48]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody | 6.97 [5.05 to 9.61] | 7.73 [5.90 to 10.13] | 4.44 [3.28 to 6.01] | 6.53 [4.74 to 9.00] | 5.45 [4.12 to 7.20] | 7.68 [5.75 to 10.28] | 5.93 [4.42 to 7.96] | 6.98 [5.58 to 8.73]
  Influenza B/Victoria Lineage | 3.45 [2.62 to 4.54] | 2.48 [1.98 to 3.12] | 1.93 [1.60 to 2.32] | 2.37 [2.01 to 2.80] | 2.40 [1.92 to 3.01] | 2.35 [1.99 to 2.78] | 2.50 [2.08 to 3.00] | 2.37 [1.94 to 2.90]
  Influenza B/Yamagata Lineage | 3.75 [2.89 to 4.88] | 3.12 [2.49 to 3.90] | 2.83 [2.31 to 3.47] | 3.62 [2.88 to 4.57] | 3.18 [2.64 to 3.81] | 3.65 [2.94 to 4.53] | 2.98 [2.46 to 3.61] | 4.05 [3.25 to 5.04]

7. Primary Outcome: GMFR of Anti-NA Antibodies at Day 29 as Measured by NAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI was calculated based on the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation.
Time Frame: Day 29
Population: PP Set consisted of all participants in the FAS who complied with injection schedule, complied with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, did not had influenza infection at baseline through Day 29, and had no major protocol deviations that impacted immune response. Here, Number analyzed signifies those who were evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 67 | 63 | 67 | 66 | 66 | 64 | 67 | 63
ratio
  Influenza A H1N1 Antibody | 1.01 [0.93 to 1.10] | 1.00 [0.96 to 1.05] | 1.42 [1.23 to 1.65] | 2.18 [1.80 to 2.63] | 1.82 [1.57 to 2.11] | 2.35 [1.92 to 2.89] | 1.75 [1.49 to 2.05] | 2.38 [1.96 to 2.90]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 67 | 63 | 67 | 66 | 66 | 64 | 66 | 63
  Influenza A H3N2 Antibody | 0.94 [0.84 to 1.05] | 1.07 [0.92 to 1.24] | 3.18 [2.41 to 4.21] | 4.61 [3.64 to 5.84] | 3.65 [2.79 to 4.79] | 6.29 [4.80 to 8.23] | 4.47 [3.43 to 5.83] | 8.01 [6.04 to 10.64]
  Influenza B/Victoria Lineage | 0.93 [0.86 to 1.01] | 0.99 [0.90 to 1.08] | 3.57 [2.95 to 4.32] | 5.78 [4.80 to 6.95] | 4.31 [3.63 to 5.10] | 6.80 [5.67 to 8.16] | 4.30 [3.64 to 5.08] | 6.49 [5.43 to 7.76]
  Influenza B/Yamagata Lineage | 1.00 [0.92 to 1.09] | 0.95 [0.86 to 1.05] | 4.21 [3.48 to 5.10] | 6.76 [5.41 to 8.46] | 4.54 [3.79 to 5.43] | 7.74 [6.35 to 9.45] | 4.87 [4.07 to 5.82] | 8.36 [6.82 to 10.24]

8. Primary Outcome: Percentage of Participants With Seroconversion as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B
Description: Seroconversion at a participant level is defined as corresponding visit titer ≥ 4*LLOQ (lower limit of quantification) if baseline is < LLOQ or a 4-fold or greater rise if baseline is ≥ LLOQ in anti-HA antibodies. When LLOQ is 1:10, seroconversion is defined as a corresponding visit titer ≥ 1:40 if baseline is < 1:10 or a 4-fold or greater rise if baseline is ≥ 1:10 in anti- HA antibodies measured by HAI assay. 95% CI was calculated using the Clopper-Pearson method.
Time Frame: Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 65 | 61 | 67 | 63 | 63 | 60 | 66 | 61
percentage of participants
  Influenza A H1N1 Antibody | 66.2 [53.35 to 77.43] | 75.4 [62.71 to 85.54] | 56.7 [44.04 to 68.78] | 74.6 [62.06 to 84.73] | 71.4 [58.65 to 82.11] | 71.7 [58.56 to 82.55] | 69.7 [57.15 to 80.41] | 67.2 [54.00 to 78.69]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody | 69.2 [56.55 to 80.09] | 73.8 [60.93 to 84.20] | 50.0 [37.43 to 62.57] | 65.1 [52.03 to 76.66] | 60.3 [47.20 to 72.43] | 76.7 [63.96 to 86.62] | 65.2 [52.42 to 76.47] | 82.0 [70.02 to 90.64]
  Influenza B/Victoria Lineage | 46.2 [33.70 to 58.97] | 19.7 [10.60 to 31.84] | 14.9 [7.40 to 25.74] | 28.6 [17.89 to 41.35] | 30.2 [19.23 to 43.02] | 25.0 [14.72 to 37.86] | 25.8 [15.78 to 38.01] | 23.0 [13.15 to 35.50]
  Influenza B/Yamagata Lineage | 47.7 [35.15 to 60.46] | 36.1 [24.16 to 49.37] | 37.3 [25.80 to 49.99] | 52.4 [39.41 to 65.12] | 41.3 [29.01 to 54.38] | 45.0 [32.12 to 58.39] | 40.9 [28.95 to 53.71] | 54.1 [40.85 to 66.94]

9. Primary Outcome: Percentage of Participants With a Change in the Day 29 Titer of at Least 2-/3-/4-Fold Rise by HAI Assay
Description: ≥ z-fold rise from baseline at participant level is defined as a ≥ z x LLOQ for participants with baseline antibody level < LLOQ, or a z-times or higher antibody level ratio in participants with baseline antibody level ≥ LLOQ. 95% CI was calculated using the Clopper-Pearson method.
Time Frame: Baseline (Day 1), Day 29
Population: PP Set consisted of all participants in the FAS who complied with injection schedule, complied with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, did not had influenza infection at baseline through Day 29, and had no major protocol deviations that impacted immune response.Number of participants analyzed signifies those who were evaluable for this outcome measure. Number analyzed signifies those who were evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 65 | 61 | 67 | 63 | 63 | 60 | 66 | 61
Percentage of Participants
  Influenza A H1N1 Antibody: ≥ 2-fold Rise from Baseline | 84.6 [73.52 to 92.37] | 93.4 [84.05 to 98.18] | 80.6 [69.11 to 89.24] | 84.1 [72.74 to 92.12] | 92.1 [82.44 to 97.37] | 93.3 [83.30 to 98.15] | 92.4 [83.20 to 97.49] | 95.1 [86.29 to 98.97]
  Influenza A H1N1 Antibody: ≥ 3-fold Rise from Baseline | 67.7 [54.95 to 78.77] | 77.0 [64.50 to 86.85] | 56.7 [44.04 to 68.78] | 74.6 [62.06 to 84.73] | 71.4 [58.65 to 82.11] | 71.7 [58.56 to 82.55] | 69.7 [57.15 to 80.41] | 68.9 [55.71 to 80.10]
  Influenza A H1N1 Antibody: ≥ 4-fold Rise from Baseline | 66.2 [53.35 to 77.43] | 75.4 [62.71 to 85.54] | 56.7 [44.04 to 68.78] | 74.6 [62.06 to 84.73] | 71.4 [58.65 to 82.11] | 71.7 [58.56 to 82.55] | 69.7 [57.15 to 80.41] | 67.2 [54.00 to 78.69]
  Influenza A H3N2 Antibody: ≥ 2-fold Rise from Baseline: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody: ≥ 2-fold Rise from Baseline | 87.7 [77.18 to 94.53] | 96.7 [88.65 to 99.60] | 80.3 [68.68 to 89.07] | 90.5 [80.41 to 96.42] | 88.9 [78.44 to 95.41] | 91.7 [81.61 to 97.24] | 92.4 [83.20 to 97.49] | 98.4 [91.20 to 99.96]
  Influenza A H3N2 Antibody: ≥ 3-fold Rise from Baseline: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody: ≥ 3-fold Rise from Baseline | 69.2 [56.55 to 80.09] | 75.4 [62.71 to 85.54] | 51.5 [38.88 to 64.01] | 65.1 [52.03 to 76.66] | 60.3 [47.20 to 72.43] | 76.7 [63.96 to 86.62] | 65.2 [52.42 to 76.47] | 82.0 [70.02 to 90.64]
  Influenza A H3N2 Antibody: ≥ 4-fold Rise from Baseline: number analyzed (Participants) | 65 | 61 | 66 | 63 | 63 | 60 | 66 | 61
  Influenza A H3N2 Antibody: ≥ 4-fold Rise from Baseline | 69.2 [56.55 to 80.09] | 73.8 [60.93 to 84.20] | 50.0 [37.43 to 62.57] | 65.1 [52.03 to 76.66] | 60.3 [47.20 to 72.43] | 76.7 [63.96 to 86.62] | 65.2 [52.42 to 76.47] | 82.0 [70.02 to 90.64]
  Influenza B/Victoria Lineage: ≥ 2-fold Rise from Baseline | 78.5 [66.51 to 87.69] | 65.6 [52.31 to 77.27] | 46.3 [34.00 to 58.88] | 68.3 [55.31 to 79.42] | 66.7 [53.66 to 78.05] | 71.7 [58.56 to 82.55] | 71.2 [58.75 to 81.70] | 68.9 [55.71 to 80.10]
  Influenza B/Victoria Lineage: ≥ 3-fold Rise from Baseline | 47.7 [35.15 to 60.46] | 19.7 [10.60 to 31.84] | 14.9 [7.40 to 25.74] | 28.6 [17.89 to 41.35] | 30.2 [19.23 to 43.02] | 25.0 [14.72 to 37.86] | 25.8 [15.78 to 38.01] | 23.0 [13.15 to 35.50]
  Influenza B/Victoria Lineage: ≥ 4-fold Rise from Baseline | 46.2 [33.70 to 58.97] | 19.7 [10.60 to 31.84] | 14.9 [7.40 to 25.74] | 28.6 [17.89 to 41.35] | 30.2 [19.23 to 43.02] | 25.0 [14.72 to 37.86] | 25.8 [15.78 to 38.01] | 23.0 [13.15 to 35.50]
  Influenza B/Yamagata Lineage: ≥ 2-fold Rise from Baseline | 75.4 [63.13 to 85.23] | 85.2 [73.83 to 93.02] | 77.6 [65.78 to 86.89] | 84.1 [72.74 to 92.12] | 87.3 [76.50 to 94.35] | 93.3 [83.30 to 98.15] | 87.9 [77.51 to 94.62] | 93.4 [84.05 to 98.18]
  Influenza B/Yamagata Lineage: ≥ 3-fold Rise from Baseline | 47.7 [35.15 to 60.46] | 36.1 [24.16 to 49.37] | 37.3 [25.80 to 49.99] | 52.4 [39.41 to 65.12] | 41.3 [29.01 to 54.38] | 45.0 [32.12 to 58.39] | 40.9 [28.95 to 53.71] | 54.1 [40.85 to 66.94]
  Influenza B/Yamagata Lineage: ≥ 4-fold Rise from Baseline | 47.7 [35.15 to 60.46] | 36.1 [24.16 to 49.37] | 37.3 [25.80 to 49.99] | 52.4 [39.41 to 65.12] | 41.3 [29.01 to 54.38] | 45.0 [32.12 to 58.39] | 40.9 [28.95 to 53.71] | 54.1 [40.85 to 66.94]

10. Secondary Outcome: GMT of Anti-HA or Anti-NA Antibodies at Days 8 and 181 as Measured by HAI and NAI Assays for Vaccine-Matched Seasonal Influenza A and B Strains
Description: as for outcome 5
Time Frame: Days 8 and 181
Population: PP Set consisted of all participants in the FAS who comply with injection schedule, comply with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, do not have influenza infection at baseline through Day 29, and have no major protocol deviations that impact immune response. Number of participants analyzed signifies those who were evaluable for this outcome measure and number analyzed signifies those who were evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 66 | 63 | 67 | 66 | 66 | 64 | 67 | 63
titer
  Day 8: Influenza A H1N1 Antibody (titer) by HAI Assay: number analyzed (Participants) | 59 | 60 | 61 | 59 | 62 | 58 | 63 | 60
  Day 8: Influenza A H1N1 Antibody (titer) by HAI Assay | 348.67 [236.32 to 514.44] | 242.49 [181.00 to 324.88] | 167.43 [122.81 to 228.25] | 207.90 [151.25 to 285.77] | 195.65 [141.71 to 270.11] | 186.93 [136.89 to 255.26] | 281.89 [212.63 to 373.72] | 344.86 [256.99 to 462.78]
  Day 181: Influenza A H1N1 Antibody (titer) by HAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza A H1N1 Antibody (titer) by HAI Assay | 203.10 [145.63 to 283.25] | 170.30 [129.94 to 223.20] | 138.97 [101.24 to 190.77] | 171.47 [124.45 to 236.24] | 141.74 [103.95 to 193.27] | 120.48 [84.40 to 171.97] | 149.60 [113.99 to 196.33] | 164.66 [121.59 to 222.99]
  Day 8: Influenza A H3N2 Antibody (titer) by HAI Assay: number analyzed (Participants) | 59 | 60 | 61 | 59 | 62 | 58 | 63 | 60
  Day 8: Influenza A H3N2 Antibody (titer) by HAI Assay | 193.05 [140.03 to 266.14] | 164.69 [123.53 to 219.55] | 151.14 [112.49 to 203.09] | 121.39 [88.43 to 166.65] | 139.91 [101.30 to 193.22] | 138.63 [97.30 to 197.50] | 190.79 [146.44 to 248.58] | 181.63 [134.14 to 245.94]
  Day 181: Influenza A H3N2 Antibody (titer) by HAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza A H3N2 Antibody (titer) by HAI Assay | 178.85 [126.64 to 252.58] | 131.90 [97.43 to 178.57] | 149.90 [111.76 to 201.04] | 116.43 [88.30 to 153.51] | 134.16 [97.23 to 185.12] | 111.81 [78.03 to 160.20] | 146.30 [112.22 to 190.74] | 131.15 [98.53 to 174.58]
  Day 8: Influenza B/Victoria Lineage (titer) by HAI Assay: number analyzed (Participants) | 59 | 60 | 61 | 59 | 62 | 58 | 63 | 60
  Day 8: Influenza B/Victoria Lineage (titer) by HAI Assay | 140.58 [106.39 to 185.76] | 80.91 [60.90 to 107.49] | 93.28 [73.73 to 117.99] | 83.35 [63.73 to 109.00] | 114.40 [91.42 to 143.16] | 101.00 [79.71 to 127.98] | 100.25 [82.12 to 122.40] | 91.30 [71.16 to 117.13]
  Day 181: Influenza B/Victoria Lineage (titer) by HAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Victoria Lineage (titer) by HAI Assay | 98.26 [73.80 to 130.81] | 64.82 [49.01 to 85.73] | 83.56 [65.97 to 105.82] | 80.49 [61.62 to 105.14] | 91.80 [72.47 to 116.28] | 74.64 [56.65 to 98.34] | 63.97 [50.20 to 81.52] | 55.26 [42.76 to 71.41]
  Day 8: Influenza B/Yamagata Lineage (titer) by HAI Assay: number analyzed (Participants) | 59 | 60 | 61 | 59 | 62 | 57 | 63 | 60
  Day 8: Influenza B/Yamagata Lineage (titer) by HAI Assay | 250.04 [195.63 to 319.58] | 188.07 [141.60 to 249.80] | 138.81 [111.32 to 173.07] | 171.63 [132.14 to 222.91] | 195.70 [153.33 to 249.78] | 227.71 [181.02 to 286.45] | 216.55 [176.59 to 265.56] | 209.90 [162.24 to 271.56]
  Day 181: Influenza B/Yamagata Lineage (titer) by HAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Yamagata Lineage (titer) by HAI Assay | 134.94 [103.17 to 176.51] | 104.47 [82.63 to 132.09] | 90.12 [69.17 to 117.42] | 113.17 [87.90 to 145.70] | 105.33 [84.91 to 130.68] | 113.74 [88.60 to 146.02] | 106.39 [86.72 to 130.52] | 93.22 [72.19 to 120.38]
  Day 8: Influenza A H1N1 Antibody (titer) by NAI Assay: number analyzed (Participants) | 66 | 63 | 67 | 65 | 66 | 64 | 67 | 63
  Day 8: Influenza A H1N1 Antibody (titer) by NAI Assay | 109.63 [92.53 to 129.89] | 96.45 [86.45 to 107.62] | 119.76 [102.45 to 140.00] | 145.36 [119.15 to 177.33] | 124.35 [108.21 to 142.90] | 136.01 [114.31 to 161.83] | 114.91 [100.62 to 131.23] | 184.60 [148.17 to 229.99]
  Day 181: Influenza A H1N1 Antibody (titer) by NAI Assay: number analyzed (Participants) | 59 | 62 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza A H1N1 Antibody (titer) by NAI Assay | 104.82 [88.93 to 123.55] | 93.55 [85.29 to 102.62] | 136.01 [112.81 to 163.97] | 149.29 [118.89 to 187.46] | 151.44 [125.37 to 182.92] | 126.99 [108.93 to 148.05] | 135.30 [114.76 to 159.51] | 161.83 [130.05 to 201.37]
  Day 8: Influenza A H3N2 Antibody (titer) by NAI Assay | 26.70 [20.25 to 35.21] | 19.59 [15.71 to 24.42] | 55.15 [39.90 to 76.24] | 64.20 [44.15 to 93.35] | 62.87 [45.00 to 87.83] | 74.58 [51.72 to 107.55] | 73.44 [53.46 to 100.89] | 79.31 [57.39 to 109.59]
  Day 181: Influenza A H3N2 Antibody (titer) by NAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 59 | 62 | 61
  Day 181: Influenza A H3N2 Antibody (titer) by NAI Assay | 21.34 [16.79 to 27.12] | 19.13 [15.27 to 23.97] | 50.91 [37.88 to 68.41] | 50.43 [35.78 to 71.07] | 50.86 [35.48 to 72.91] | 64.15 [46.15 to 89.18] | 69.34 [49.33 to 97.47] | 64.08 [45.54 to 90.17]
  Day 8: Influenza B/Victoria Lineage (titer) by NAI Assay: number analyzed (Participants) | 66 | 63 | 67 | 65 | 66 | 64 | 67 | 63
  Day 8: Influenza B/Victoria Lineage (titer) by NAI Assay | 73.55 [63.06 to 85.79] | 80.00 [67.77 to 94.44] | 209.38 [176.83 to 247.92] | 281.56 [226.25 to 350.40] | 238.47 [196.00 to 290.15] | 330.57 [267.90 to 407.90] | 282.64 [238.72 to 334.64] | 365.16 [293.96 to 453.61]
  Day 181: Influenza B/Victoria Lineage (titer) by NAI Assay: number analyzed (Participants) | 59 | 62 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Victoria Lineage (titer) by NAI Assay | 82.87 [69.08 to 99.41] | 79.11 [67.14 to 93.21] | 161.64 [136.79 to 191.24] | 236.98 [194.79 to 288.30] | 195.04 [161.84 to 235.06] | 251.07 [205.54 to 306.67] | 182.97 [150.40 to 222.60] | 214.99 [173.21 to 266.86]
  Day 8: Influenza B/Yamagata Lineage (titer) by NAI Assay | 208.04 [162.96 to 265.59] | 220.14 [180.17 to 268.96] | 640.00 [546.19 to 749.92] | 914.65 [749.75 to 1115.83] | 823.47 [696.04 to 974.22] | 1064.75 [879.83 to 1288.55] | 828.90 [698.48 to 983.68] | 1085.27 [873.94 to 1347.70]
  Day 181: Influenza B/Yamagata Lineage (titer) by NAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Yamagata Lineage (titer) by NAI Assay | 193.09 [150.62 to 247.53] | 212.57 [173.00 to 261.18] | 414.99 [343.55 to 501.28] | 625.38 [517.53 to 755.70] | 536.70 [450.77 to 639.00] | 693.91 [561.72 to 857.20] | 529.22 [436.91 to 641.05] | 604.65 [489.74 to 746.53]

11. Secondary Outcome: GMFR of Anti-HA or Anti-NA Antibodies at Days 8 and 181 as Measured by HAI and NAI Assays for Vaccine-Matched Seasonal Influenza A and B Strains
Description: as for outcome 7
Time Frame: Days 8 and 181
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
Number analyzed (Participants) | 66 | 63 | 67 | 66 | 66 | 64 | 67 | 63
ratio
  Day 8: Influenza A H1N1 Antibody (titer) by HAI Assay: number analyzed (Participants) | 57 | 58 | 61 | 56 | 59 | 54 | 62 | 59
  Day 8: Influenza A H1N1 Antibody (titer) by HAI Assay | 4.37 [2.79 to 6.87] | 4.32 [3.18 to 5.89] | 2.78 [2.04 to 3.79] | 3.97 [2.89 to 5.47] | 3.18 [2.24 to 4.54] | 4.16 [3.00 to 5.78] | 4.65 [3.43 to 6.30] | 4.32 [3.11 to 6.00]
  Day 181: Influenza A H1N1 Antibody (titer) by HAI Assay: number analyzed (Participants) | 57 | 60 | 64 | 57 | 60 | 57 | 61 | 60
  Day 181: Influenza A H1N1 Antibody (titer) by HAI Assay | 2.71 [1.88 to 3.90] | 3.07 [2.25 to 4.19] | 2.24 [1.59 to 3.16] | 3.34 [2.30 to 4.85] | 2.64 [1.88 to 3.70] | 2.63 [1.91 to 3.63] | 2.36 [1.82 to 3.06] | 2.08 [1.55 to 2.81]
  Day 8: Influenza A H3N2 Antibody (titer) by HAI Assay: number analyzed (Participants) | 57 | 58 | 61 | 56 | 59 | 54 | 62 | 59
  Day 8: Influenza A H3N2 Antibody (titer) by HAI Assay | 3.25 [2.33 to 4.54] | 3.84 [2.79 to 5.27] | 2.78 [2.12 to 3.64] | 3.22 [2.34 to 4.43] | 3.58 [2.68 to 4.78] | 3.75 [2.79 to 5.05] | 4.02 [2.95 to 5.49] | 4.07 [3.07 to 5.40]
  Day 181: Influenza A H3N2 Antibody (titer) by HAI Assay: number analyzed (Participants) | 57 | 60 | 64 | 57 | 60 | 57 | 61 | 60
  Day 181: Influenza A H3N2 Antibody (titer) by HAI Assay | 3.37 [2.44 to 4.67] | 3.29 [2.49 to 4.34] | 2.69 [2.04 to 3.55] | 3.01 [2.27 to 3.98] | 3.65 [2.71 to 4.92] | 3.46 [2.64 to 4.52] | 2.80 [2.11 to 3.71] | 3.12 [2.50 to 3.90]
  Day 8: Influenza B/Victoria Lineage (titer) by HAI Assay: number analyzed (Participants) | 57 | 58 | 61 | 56 | 59 | 54 | 62 | 59
  Day 8: Influenza B/Victoria Lineage (titer) by HAI Assay | 2.92 [2.08 to 4.09] | 2.25 [1.75 to 2.91] | 2.28 [1.86 to 2.80] | 2.31 [1.89 to 2.81] | 2.55 [2.04 to 3.18] | 2.69 [2.12 to 3.42] | 2.83 [2.21 to 3.63] | 2.73 [2.19 to 3.41]
  Day 181: Influenza B/Victoria Lineage (titer) by HAI Assay: number analyzed (Participants) | 57 | 60 | 64 | 57 | 60 | 57 | 61 | 60
  Day 181: Influenza B/Victoria Lineage (titer) by HAI Assay | 2.13 [1.67 to 2.71] | 1.88 [1.45 to 2.43] | 1.83 [1.47 to 2.26] | 2.05 [1.67 to 2.53] | 2.14 [1.70 to 2.70] | 2.03 [1.71 to 2.40] | 1.78 [1.51 to 2.08] | 1.79 [1.45 to 2.22]
  Day 8: Influenza B/Yamagata Lineage (titer) by HAI Assay: number analyzed (Participants) | 57 | 58 | 61 | 56 | 59 | 53 | 62 | 59
  Day 8: Influenza B/Yamagata Lineage (titer) by HAI Assay | 3.03 [2.17 to 4.22] | 2.31 [1.76 to 3.03] | 2.17 [1.77 to 2.65] | 2.73 [2.06 to 3.60] | 2.52 [1.94 to 3.26] | 3.12 [2.38 to 4.10] | 2.68 [2.17 to 3.30] | 3.41 [2.62 to 4.44]
  Day 181: Influenza B/Yamagata Lineage (titer) by HAI Assay: number analyzed (Participants) | 57 | 60 | 64 | 57 | 60 | 57 | 61 | 60
  Day 181: Influenza B/Yamagata Lineage (titer) by HAI Assay | 1.62 [1.25 to 2.10] | 1.36 [1.06 to 1.74] | 1.36 [1.05 to 1.76] | 1.67 [1.35 to 2.06] | 1.45 [1.16 to 1.80] | 1.57 [1.31 to 1.88] | 1.26 [1.05 to 1.51] | 1.53 [1.22 to 1.92]
  Day 8: Influenza A H1N1 Antibody (titer) by NAI Assay: number analyzed (Participants) | 66 | 63 | 67 | 65 | 66 | 64 | 67 | 63
  Day 8: Influenza A H1N1 Antibody (titer) by NAI Assay | 1.07 [0.96 to 1.18] | 0.99 [0.94 to 1.04] | 1.04 [0.98 to 1.10] | 1.44 [1.26 to 1.64] | 1.16 [1.08 to 1.24] | 1.61 [1.37 to 1.90] | 1.18 [1.09 to 1.28] | 1.64 [1.39 to 1.93]
  Day 181: Influenza A H1N1 Antibody (titer) by NAI Assay: number analyzed (Participants) | 59 | 62 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza A H1N1 Antibody (titer) by NAI Assay | 1.00 [0.94 to 1.07] | 0.97 [0.92 to 1.02] | 1.20 [1.07 to 1.36] | 1.52 [1.26 to 1.82] | 1.39 [1.22 to 1.58] | 1.50 [1.30 to 1.73] | 1.43 [1.25 to 1.64] | 1.47 [1.28 to 1.69]
  Day 8: Influenza A H3N2 Antibody (titer) by NAI Assay | 1.21 [1.01 to 1.46] | 0.99 [0.90 to 1.09] | 2.54 [1.97 to 3.26] | 2.81 [2.17 to 3.64] | 2.89 [2.20 to 3.78] | 3.67 [2.69 to 5.01] | 3.57 [2.72 to 4.69] | 4.57 [3.32 to 6.28]
  Day 181: Influenza A H3N2 Antibody (titer) by NAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 59 | 62 | 61
  Day 181: Influenza A H3N2 Antibody (titer) by NAI Assay | 1.03 [0.85 to 1.24] | 0.98 [0.85 to 1.14] | 2.28 [1.80 to 2.87] | 2.33 [1.75 to 3.10] | 2.27 [1.77 to 2.92] | 3.20 [2.46 to 4.16] | 3.43 [2.45 to 4.81] | 3.65 [2.68 to 4.96]
  Day 8: Influenza B/Victoria Lineage (titer) by NAI Assay: number analyzed (Participants) | 66 | 63 | 67 | 65 | 66 | 64 | 67 | 63
  Day 8: Influenza B/Victoria Lineage (titer) by NAI Assay | 0.97 [0.88 to 1.06] | 1.01 [0.92 to 1.11] | 2.78 [2.27 to 3.41] | 3.96 [3.18 to 4.93] | 3.24 [2.65 to 3.97] | 4.71 [3.79 to 5.85] | 3.84 [3.15 to 4.67] | 5.04 [3.95 to 6.43]
  Day 181: Influenza B/Victoria Lineage (titer) by NAI Assay: number analyzed (Participants) | 59 | 62 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Victoria Lineage (titer) by NAI Assay | 1.06 [0.93 to 1.21] | 1.00 [0.92 to 1.08] | 2.16 [1.79 to 2.60] | 3.36 [2.78 to 4.07] | 2.69 [2.33 to 3.12] | 3.52 [2.89 to 4.30] | 2.45 [2.12 to 2.82] | 3.01 [2.48 to 3.66]
  Day 8: Influenza B/Yamagata Lineage (titer) by NAI Assay | 1.12 [0.97 to 1.30] | 0.97 [0.87 to 1.08] | 3.22 [2.64 to 3.92] | 4.78 [3.72 to 6.14] | 3.92 [3.13 to 4.91] | 5.72 [4.45 to 7.35] | 4.04 [3.27 to 4.99] | 6.35 [4.76 to 8.46]
  Day 181: Influenza B/Yamagata Lineage (titer) by NAI Assay: number analyzed (Participants) | 59 | 61 | 64 | 60 | 63 | 60 | 62 | 61
  Day 181: Influenza B/Yamagata Lineage (titer) by NAI Assay | 1.02 [0.89 to 1.18] | 0.96 [0.85 to 1.07] | 2.11 [1.81 to 2.47] | 3.44 [2.75 to 4.31] | 2.63 [2.25 to 3.09] | 3.65 [3.03 to 4.39] | 2.53 [2.17 to 2.95] | 3.61 [2.90 to 4.50]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 181
Description: Safety Analysis Set consisted of all randomly assigned participants who received the investigational product. Participants were included in the vaccination group corresponding to the study injection they actually received. Note, not all solicited ARs were considered AEs. The Investigator reviewed whether the solicited AR was also to be recorded as an AE. All cause mortality was based on the randomized set.
Arm/Group | Flublok | mRNA-1010 | mRNA-1030 Dose Level A | mRNA-1020 Dose Level A | mRNA-1030 Dose Level B | mRNA-1020 Dose Level B | mRNA-1030 Dose Level C | mRNA-1020 Dose Level C
All-Cause Mortality (participants affected / at risk) | 1/72 | 0/71 | 0/71 | 0/72 | 0/72 | 0/71 | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/71 | 1/71 | 1/71 | 1/71 | 1/72 | 0/67 | 2/72 | 4/70
Other Adverse Events (participants affected / at risk) | 58/71 | 67/71 | 62/71 | 66/71 | 63/72 | 62/67 | 70/72 | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok (N=71) | mRNA-1010 (N=71) | mRNA-1030 Dose Level A (N=71) | mRNA-1020 Dose Level A (N=71) | mRNA-1030 Dose Level B (N=72) | mRNA-1020 Dose Level B (N=67) | mRNA-1030 Dose Level C (N=72) | mRNA-1020 Dose Level C (N=70)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal wall cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok (N=71) | mRNA-1010 (N=71) | mRNA-1030 Dose Level A (N=71) | mRNA-1020 Dose Level A (N=71) | mRNA-1030 Dose Level B (N=72) | mRNA-1020 Dose Level B (N=67) | mRNA-1030 Dose Level C (N=72) | mRNA-1020 Dose Level C (N=70)
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 2 | 1 | 6 | 7 | 4 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 5 | 2 | 3 | 1 | 2
Rhinovirus infection (Infections and infestations) | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 16 | 46 | 30 | 42 | 34 | 48 | 49 | 50
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 23 | 13 | 31 | 34 | 37 | 40 | 44
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 18 | 44 | 33 | 46 | 46 | 49 | 54 | 56
Injection site pain (General disorders) | 35 | 61 | 59 | 59 | 55 | 57 | 67 | 67
Injection site lymphadenopathy (General disorders) | 10 | 25 | 18 | 16 | 20 | 20 | 28 | 27
Injection site erythema (General disorders) | 2 | 3 | 1 | 3 | 2 | 5 | 6 | 12
Injection site induration (General disorders) | 2 | 5 | 4 | 4 | 5 | 10 | 8 | 15
Haemoglobin decreased (Investigations) | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 12 | 9 | 10 | 15 | 10 | 16 | 13
Chills (General disorders) | 8 | 30 | 15 | 23 | 30 | 35 | 41 | 39
Pyrexia (General disorders) | 0 | 10 | 2 | 3 | 8 | 10 | 10 | 12
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 38 | 20 | 40 | 42 | 46 | 51 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05333289/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT05333289/SAP_001.pdf